CLINICAL TRIAL: NCT00442104
Title: An Open-label Clinical Study to Evaluate the Safety and Antiepileptic Activity of Ganaxolone in Treatment of Patients Diagnosed With Infantile Spasms.
Brief Title: Open-label Extension to Protocol 1042-0500
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Marinus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1042-0501; Amend 5 (ROW); Amend 6 (US)
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Results first posted 2023-06-02 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Infantile Spasms
Keywords: infantile spasms; anticonvulsant; pediatric epilepsy; West Syndrome; epileptic spasms
MeSH Terms: conditions — Spasms, Infantile | interventions — ganaxolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ganaxolone (Experimental)
  Interventions: Drug: Ganaxolone

INTERVENTIONS:
Drug: Ganaxolone

SUMMARY:
To allow open-label extension to patients who have completed Protocol 1042-0500

DETAILED DESCRIPTION:
Patient should have completed all scheduled clinical study visits in the double blind, controlled trial (Protocol 1042-0500) and have been deemed eligible (had a response to treatment) by the Investigator. Male or female, with a diagnosis of IS with a video EEG (vEEG) recording confirming the diagnosis.

There will be a total of 14 visits over 99(+or-1)week. A 24-hr vEEG is only required if the subject has been spasm-free for more than 24-hrs.

ELIGIBILITY:
Inclusion Criteria:

* Have completed all scheduled clinical study visits in the previous Protocol 1042 0500 and have been deemed eligible (no SAEs thought to be drug related and had a response to treatment) by the Investigator.
* Be diagnosed with IS regardless of etiology. Diagnostic Criteria: Seizures consisting of single or repetitive short muscular contractions leading to flexion or extension. Spasms may be characterized as tonic or myoclonic contractions, may occur singly or in clusters, and typically occur bilaterally and symmetrically. The EEG pattern must be consistent with the diagnosis of IS (hypsarrhythmia, modified hypsarrhythmia, multifocal spike wave discharges, etc).
* Have a 24 hour vEEG recording confirming the diagnosis of IS.
* Have had a magnetic resonance imaging (MRI) performed to determine any possible causes of IS.
* Have been previously treated with 3 AEDs or fewer.
* Have a parent/guardian who is properly informed of the nature and potential risks and benefits of the clinical study, is willing and capable of complying with all clinical study procedures, and has given informed consent in writing prior to entering the clinical study.

Exclusion Criteria:

* Current treatment with more than 2 concomitant AEDs.
* Have an active CNS infection, demyelinating disease, degenerative neurological disease, or CNS disease deemed progressive (with the exception of tuberous sclerosis) as evaluated by brain MRI.
* Have any disease or condition (medical or surgical) at Screening that might compromise the hematologic, cardiovascular, pulmonary, renal, GI, or hepatic systems; or other conditions that might interfere with the absorption, distribution, metabolism, or excretion of the investigational product, or would place the subject at increased risk.
* Aspartate transaminase (AST), alanine transaminase (ALT), or total bilirubin greater than 4 times the upper limit of laboratory normal or any clinical laboratory value deemed clinically significant by the Investigator.
* History of recurrent status epilepticus.
* Have been exposed to any other investigational drug within 30 days prior to enrollment.

Ages: 4 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Mattel Children's Hospital at UCLA, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Miami Children's Hospital, The Brain Institute, Miami, Florida
  - Child Neurology Center of Nrothwest Florida, P.A., Pensacola, Florida
  - University of Chicago Comer Children's Hospital, Chicago, Illinois
  - Minnesota Epilepsy Group, P.A., Saint Paul, Minnesota
  - Montefiore Medical Center- Albert Einstein College of Medicine, The Bronx, New York
  - Le Bonheur Children's Medical Center, Memphis, Tennessee
  - Dallas Pediatric Neurology Associates, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Virginia Commonwealth University Health Systems, Richmond, Virginia
  - Children's Hospital and Regional Medical Center, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed the previous double-blind controlled trial (Protocol 1042-0500, NCT00441896) were enrolled in this study. No separate analysis was performed to report results by doses.
Groups:
- Ganaxolone: Participants were administered a maximum dose of 54 milligrams per kilogram (mg/kg)/day ganaxolone oral suspension. The investigator could adjust (increase or decrease) the dose of ganaxolone by 3 mg/kg three times a day (total daily dose adjustment = 9 mg/kg) until the optimal dose for efficacy and tolerability was achieved
Period: Overall Study
Arm/Group | Ganaxolone
Started | 54
Completed | 7
Not Completed | 47
Not completed — Adverse Event | 5
Not completed — Death | 2
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 5
Not completed — Insufficient Clinical Response | 10
Not completed — Other | 21
Not completed — Discretion of the Investigator/Sponsor | 1

BASELINE CHARACTERISTICS:
Groups:
- Ganaxolone: Participants were administered a maximum dose of 54 mg/kg/day ganaxolone oral suspension. The investigator could adjust (increase or decrease) the dose of ganaxolone by 3 mg/kg t.i.d. (total daily dose adjustment = 9 mg/kg) until the optimal dose for efficacy and tolerability was achieved.
Arm/Group | Ganaxolone
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: months] | 13.4 (6.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 33
  More than one race | 0
  Unknown or Not Reported | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Were Free of Spasms
Description: Clinical spasms were determined by video-electroencephalography (VEEG). The number of participants with spasm-free duration have been presented.
Time Frame: Weeks 4 through Week 96
Population: ITT Population included all participants who received at least 1 dose of open-label study medication. Only those participants with data available at the indicated time point were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ganaxolone
Number analyzed (Participants) | 7
percentage of participants | 100 [59.0 to 100.0]

2. Secondary Outcome: Change From Baseline in Frequency of Spasm Clusters
Description: Infantile spasms that come one after another in a cluster and lasts several minutes are called Spasm Clusters. Spasm clusters were determined by a 24-hour video-electroencephalography (vEEG). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Baseline was defined as the Day 0 assessment prior to ganaxolone dosing in Protocol 1042-0500.
Time Frame: Baseline and Week 4 through Week 32
Population: ITT Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: Spasm clusters per day
Arm/Group | Ganaxolone
Number analyzed (Participants) | 40
Spasm clusters per day
  Spasm Clusters - Week 4 | -2.9 (7.94)
  Spasm Clusters - Week 8: number analyzed (Participants) | 32
  Spasm Clusters - Week 8 | -4.1 (8.35)
  Spasm Clusters - Week 14: number analyzed (Participants) | 31
  Spasm Clusters - Week 14 | -4.1 (9.12)
  Spasm Clusters - Week 20: number analyzed (Participants) | 30
  Spasm Clusters - Week 20 | -5.8 (8.58)
  Spasm Clusters - Week 26: number analyzed (Participants) | 27
  Spasm Clusters - Week 26 | -5.6 (7.98)
  Spasm Clusters - Week 32: number analyzed (Participants) | 23
  Spasm Clusters - Week 32 | -5.3 (9.96)

3. Secondary Outcome: Change From Baseline in Frequency of Individual Spasm
Description: Individual Spasm are seizures that may last only a second or two and were determined by a 24-hour video-electroencephalography (vEEG). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Baseline was defined as the Day 0 assessment prior to ganaxolone dosing in Protocol 1042-0500.
Time Frame: Baseline and Week 4 through Week 32
Population: ITT Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: Individual spasms per day
Arm/Group | Ganaxolone
Number analyzed (Participants) | 39
Individual spasms per day
  Individual Spasms - Week 4 | -6.8 (40.70)
  Individual Spasms - Week 8: number analyzed (Participants) | 31
  Individual Spasms - Week 8 | -17.4 (31.28)
  Individual Spasms - Week 14: number analyzed (Participants) | 30
  Individual Spasms - Week 14 | -20.8 (31.21)
  Individual Spasms - Week 20: number analyzed (Participants) | 29
  Individual Spasms - Week 20 | -15.8 (52.46)
  Individual Spasms - Week 26: number analyzed (Participants) | 26
  Individual Spasms - Week 26 | -19.9 (39.27)
  Individual Spasms - Week 32: number analyzed (Participants) | 21
  Individual Spasms - Week 32 | -17.7 (36.35)

4. Secondary Outcome: Number of Participants With Change in Clinical Status on Caregiver's Global Assessment
Description: Caregiver global assessment of seizure severity and response to treatment rated the participants' based on 7 clinical factors: seizure frequency, duration, and intensity; adverse experiences; social, intellectual, and motor functioning. Using a 7-point scale ([1] marked improvement, [2] moderate improvement, [3] slight improvement, [4] no change from baseline, [5] slight worsening, [6] moderate worsening, or [7] marked worsening). Higher score indicated worse symptoms. The assessment compared the participants' current status to their condition prior to initiating study medication.
Time Frame: Week 4 through Week 32
Population: ITT population. Only those participants with data available at the indicated time point were analyzed.
Measure: Number; unit: participants
Arm/Group | Ganaxolone
Number analyzed (Participants) | 45
participants
  Caregiver's- Week 4 - Marked Improvement | 11
  Caregiver's - Week 4 - Moderate Improvement | 11
  Caregiver's -Week 4 - Slight Improvement | 16
  Caregiver's- Week 4 - No change from Baseline | 6
  Caregiver's - Week 4 - Moderate Worsening | 0
  Caregiver's - Week 4 - Slight Worsening | 1
  Caregiver's - Week 4 - Marked Worsening | 0
  Caregiver's - Week 8 - Marked Improvement: number analyzed (Participants) | 40
  Caregiver's - Week 8 - Marked Improvement | 7
  Caregiver's- Week 8 - Moderate Improvement: number analyzed (Participants) | 40
  Caregiver's- Week 8 - Moderate Improvement | 12
  Caregiver's -Week 8 - Slight Improvement: number analyzed (Participants) | 40
  Caregiver's -Week 8 - Slight Improvement | 18
  Caregiver's- Week 8 - No change from Baseline: number analyzed (Participants) | 40
  Caregiver's- Week 8 - No change from Baseline | 1
  Caregiver's - Week 8 - Slight Worsening: number analyzed (Participants) | 40
  Caregiver's - Week 8 - Slight Worsening | 2
  Caregiver's - Week 8 - Moderate Worsening: number analyzed (Participants) | 40
  Caregiver's - Week 8 - Moderate Worsening | 0
  Caregiver's - Week 8 - Marked Worsening: number analyzed (Participants) | 40
  Caregiver's - Week 8 - Marked Worsening | 0
  Caregiver's- Week 14 - Marked Improvement: number analyzed (Participants) | 38
  Caregiver's- Week 14 - Marked Improvement | 8
  Caregiver's - Week 14 - Moderate Improvement: number analyzed (Participants) | 38
  Caregiver's - Week 14 - Moderate Improvement | 13
  Caregiver's -Week 14 - Slight Improvement: number analyzed (Participants) | 38
  Caregiver's -Week 14 - Slight Improvement | 14
  Caregiver's - Week 14 - No change from Baseline: number analyzed (Participants) | 38
  Caregiver's - Week 14 - No change from Baseline | 2
  Caregiver's - Week 14 - Slight Worsening: number analyzed (Participants) | 38
  Caregiver's - Week 14 - Slight Worsening | 1
  Caregiver's - Week 14 - Moderate Worsening: number analyzed (Participants) | 38
  Caregiver's - Week 14 - Moderate Worsening | 0
  Caregiver's - Week 14 - Marked Worsening: number analyzed (Participants) | 38
  Caregiver's - Week 14 - Marked Worsening | 0
  Caregiver's - Week 20 - Marked Improvement: number analyzed (Participants) | 36
  Caregiver's - Week 20 - Marked Improvement | 9
  Caregiver's - Week 20 - Moderate Improvement: number analyzed (Participants) | 36
  Caregiver's - Week 20 - Moderate Improvement | 13
  Caregiver's -Week 20 - Slight Improvement: number analyzed (Participants) | 36
  Caregiver's -Week 20 - Slight Improvement | 10
  Caregiver's- Week 20 - No change from Baseline: number analyzed (Participants) | 36
  Caregiver's- Week 20 - No change from Baseline | 3
  Caregiver's- Week 20 - Slight Worsening: number analyzed (Participants) | 36
  Caregiver's- Week 20 - Slight Worsening | 1
  Caregiver's - Week 20 - Moderate Worsening: number analyzed (Participants) | 36
  Caregiver's - Week 20 - Moderate Worsening | 0
  Caregiver's - Week 20 - Marked Worsening: number analyzed (Participants) | 36
  Caregiver's - Week 20 - Marked Worsening | 0
  Caregiver's- Week 26 - Marked Improvement: number analyzed (Participants) | 31
  Caregiver's- Week 26 - Marked Improvement | 9
  Caregiver's- Week 26 - Moderate Improvement: number analyzed (Participants) | 31
  Caregiver's- Week 26 - Moderate Improvement | 12
  Caregiver's -Week 26 - Slight Improvement: number analyzed (Participants) | 31
  Caregiver's -Week 26 - Slight Improvement | 7
  Caregiver's - Week 26 - No change from Baseline: number analyzed (Participants) | 31
  Caregiver's - Week 26 - No change from Baseline | 3
  Caregiver's - Week 26 - Slight Worsening: number analyzed (Participants) | 31
  Caregiver's - Week 26 - Slight Worsening | 0
  Caregiver's - Week 26 - Moderate Worsening: number analyzed (Participants) | 31
  Caregiver's - Week 26 - Moderate Worsening | 0
  Caregiver's - Week 26 - Marked Worsening: number analyzed (Participants) | 31
  Caregiver's - Week 26 - Marked Worsening | 0
  Caregiver's - Week 32 - Marked Improvement: number analyzed (Participants) | 26
  Caregiver's - Week 32 - Marked Improvement | 8
  Caregiver's - Week 32 - Moderate Improvement: number analyzed (Participants) | 26
  Caregiver's - Week 32 - Moderate Improvement | 7
  Caregiver's-Week 32 - Slight Improvement: number analyzed (Participants) | 26
  Caregiver's-Week 32 - Slight Improvement | 8
  Caregiver's - Week 32 - No change from Baseline: number analyzed (Participants) | 26
  Caregiver's - Week 32 - No change from Baseline | 2
  Caregiver's - Week 32 - Slight Worsening: number analyzed (Participants) | 26
  Caregiver's - Week 32 - Slight Worsening | 0
  Caregiver's - Week 32 - Moderate Worsening: number analyzed (Participants) | 26
  Caregiver's - Week 32 - Moderate Worsening | 1
  Caregiver's - Week 32 - Marked Worsening: number analyzed (Participants) | 26
  Caregiver's - Week 32 - Marked Worsening | 0

5. Secondary Outcome: Number of Participants With Change in Clinical Status on the Investigator's Global Assessment
Description: The investigators rated the participants' overall clinical status based on 7 clinical factors: seizure frequency, duration, and intensity; adverse experiences; social, intellectual, and motor functioning. Using a 7-point scale ([1] marked improvement, [2] moderate improvement, [3] slight improvement, [4] no change from baseline, [5] slight worsening, [6] moderate worsening, or [7] marked worsening). Higher score indicated worse symptoms. The investigators assessed the participants' status compared to their condition prior to initiating study medication.
Time Frame: Week 4 through Week 32
Population: ITT population. Only those participants with data available at the indicated time point were analyzed.
Measure: Number; unit: participants
Arm/Group | Ganaxolone
Number analyzed (Participants) | 45
participants
  Investigator's- Week 4 - Marked Improvement | 7
  Investigator's - Week 4 - Moderate Improvement | 15
  Investigator's -Week 4 - Slight Improvement | 18
  Investigator's- Week 4 - No change from Baseline | 4
  Investigator's - Week 4 - Moderate Worsening | 1
  Investigator's - Week 4 - Slight Worsening | 0
  Investigator's - Week 4 - Marked Worsening | 0
  Investigator's - Week 8 - Marked Improvement: number analyzed (Participants) | 40
  Investigator's - Week 8 - Marked Improvement | 6
  Investigator's- Week 8 - Moderate Improvement: number analyzed (Participants) | 40
  Investigator's- Week 8 - Moderate Improvement | 12
  Investigator's -Week 8 - Slight Improvement: number analyzed (Participants) | 40
  Investigator's -Week 8 - Slight Improvement | 19
  Investigator's- Week 8 - No change from Baseline: number analyzed (Participants) | 40
  Investigator's- Week 8 - No change from Baseline | 3
  Investigator's - Week 8 - Slight Worsening: number analyzed (Participants) | 40
  Investigator's - Week 8 - Slight Worsening | 0
  Investigator's - Week 8 - Moderate Worsening: number analyzed (Participants) | 40
  Investigator's - Week 8 - Moderate Worsening | 0
  Investigator's - Week 8 - Marked Worsening: number analyzed (Participants) | 40
  Investigator's - Week 8 - Marked Worsening | 0
  Investigator's- Week 14 - Marked Improvement: number analyzed (Participants) | 38
  Investigator's- Week 14 - Marked Improvement | 6
  Investigator's - Week 14 - Moderate Improvement: number analyzed (Participants) | 38
  Investigator's - Week 14 - Moderate Improvement | 16
  Investigator's -Week 14 - Slight Improvement: number analyzed (Participants) | 38
  Investigator's -Week 14 - Slight Improvement | 15
  Investigator's - Week 14 - No change from Baseline: number analyzed (Participants) | 38
  Investigator's - Week 14 - No change from Baseline | 1
  Investigator's - Week 14 - Slight Worsening: number analyzed (Participants) | 38
  Investigator's - Week 14 - Slight Worsening | 0
  Investigator's - Week 14 - Moderate Worsening: number analyzed (Participants) | 38
  Investigator's - Week 14 - Moderate Worsening | 0
  Investigator's - Week 14 - Marked Worsening: number analyzed (Participants) | 38
  Investigator's - Week 14 - Marked Worsening | 0
  Investigator's - Week 20 - Marked Improvement: number analyzed (Participants) | 34
  Investigator's - Week 20 - Marked Improvement | 7
  Investigator's - Week 20 - Moderate Improvement: number analyzed (Participants) | 34
  Investigator's - Week 20 - Moderate Improvement | 14
  Investigator's -Week 20 - Slight Improvement: number analyzed (Participants) | 34
  Investigator's -Week 20 - Slight Improvement | 11
  Investigator's- Week 20 - No change from Baseline: number analyzed (Participants) | 34
  Investigator's- Week 20 - No change from Baseline | 1
  Investigator's- Week 20 - Slight Worsening: number analyzed (Participants) | 34
  Investigator's- Week 20 - Slight Worsening | 1
  Investigator's - Week 20 - Moderate Worsening: number analyzed (Participants) | 34
  Investigator's - Week 20 - Moderate Worsening | 0
  Investigator's - Week 20 - Marked Worsening: number analyzed (Participants) | 34
  Investigator's - Week 20 - Marked Worsening | 0
  Investigator's- Week 26 - Marked Improvement: number analyzed (Participants) | 32
  Investigator's- Week 26 - Marked Improvement | 5
  Investigator's- Week 26 - Moderate Improvement: number analyzed (Participants) | 32
  Investigator's- Week 26 - Moderate Improvement | 14
  Investigator's -Week 26 - Slight Improvement: number analyzed (Participants) | 32
  Investigator's -Week 26 - Slight Improvement | 9
  Investigator's - Week 26 - No change from Baseline: number analyzed (Participants) | 32
  Investigator's - Week 26 - No change from Baseline | 4
  Investigator's - Week 26 - Slight Worsening: number analyzed (Participants) | 32
  Investigator's - Week 26 - Slight Worsening | 0
  Investigator's - Week 26 - Moderate Worsening: number analyzed (Participants) | 32
  Investigator's - Week 26 - Moderate Worsening | 0
  Investigator's - Week 26 - Marked Worsening: number analyzed (Participants) | 32
  Investigator's - Week 26 - Marked Worsening | 0
  Investigator's - Week 32 - Marked Improvement: number analyzed (Participants) | 27
  Investigator's - Week 32 - Marked Improvement | 6
  Investigator's - Week 32 - Moderate Improvement: number analyzed (Participants) | 27
  Investigator's - Week 32 - Moderate Improvement | 9
  Investigator's -Week 32 - Slight Improvement: number analyzed (Participants) | 27
  Investigator's -Week 32 - Slight Improvement | 8
  Investigator's - Week 32 - No change from Baseline: number analyzed (Participants) | 27
  Investigator's - Week 32 - No change from Baseline | 3
  Investigator's - Week 32 - Slight Worsening: number analyzed (Participants) | 27
  Investigator's - Week 32 - Slight Worsening | 1
  Investigator's - Week 32 - Moderate Worsening: number analyzed (Participants) | 27
  Investigator's - Week 32 - Moderate Worsening | 0
  Investigator's - Week 32 - Marked Worsening: number analyzed (Participants) | 27
  Investigator's - Week 32 - Marked Worsening | 0

6. Secondary Outcome: Number of Participants With Spasm-free Durations
Description: Spasm-free duration is defined as total number of spasm-free days recorded in the spasm/seizure diary. Parents/Guardians or nursing staff maintained a spasm/seizure diary to record the number and type of seizures each day, including spasms, throughout the entire study. The number of participants with spasm-free duration of at least 24 hours have been presented.
Time Frame: Week 4 through Week 32
Population: ITT Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone
Number analyzed (Participants) | 43
Participants
  Spasm Free at Week 4 | 19
  Spasm Free at Week 8: number analyzed (Participants) | 37
  Spasm Free at Week 8 | 18
  Spasm Free at Week 14: number analyzed (Participants) | 36
  Spasm Free at Week 14 | 18
  Spasm Free at Week 20: number analyzed (Participants) | 34
  Spasm Free at Week 20 | 18
  Spasm Free at Week 26: number analyzed (Participants) | 30
  Spasm Free at Week 26 | 17
  Spasm Free at Week 32: number analyzed (Participants) | 26
  Spasm Free at Week 32 | 13

7. Secondary Outcome: Number of Participants With Absence of Spasms
Description: Absence of spasms is defined as percentage of total spasm-free days during a visit period=100%. Parents/Guardians or nursing staff maintained a spasm/seizure diary to record the number and type of seizures each day, including spasms, throughout the entire study. The participants achieving absence of spasms have been presented.
Time Frame: Week 4 through Week 32
Population: ITT Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Ganaxolone
Number analyzed (Participants) | 43
Participants
  Achieved absence of spasms at Week 4 | 2
  Achieved absence of spasms at Week 8: number analyzed (Participants) | 37
  Achieved absence of spasms at Week 8 | 3
  Achieved absence of spasms at Week 14: number analyzed (Participants) | 36
  Achieved absence of spasms at Week 14 | 3
  Achieved absence of spasms at Week 20: number analyzed (Participants) | 34
  Achieved absence of spasms at Week 20 | 4
  Achieved absence of spasms at Week 26: number analyzed (Participants) | 30
  Achieved absence of spasms at Week 26 | 5
  Achieved absence of spasms at Week 32: number analyzed (Participants) | 26
  Achieved absence of spasms at Week 32 | 1

8. Secondary Outcome: Developmental Assessment Using Denver-II Developmental Test
Description: Denver-II Developmental Test measures a child's development in several areas:Personal-Social,Fine Motor-Adaptive,Language,and Gross Motor,from birth to 6 years old.It consists of 125 items that are organized into subscales and scored as pass,fail,or refused.To evaluate a child's progress,test compares their performance to a normative sample of children of same age.For each item,age at which 90% of children in normative sample pass it is determined.Derived score for each subscale is sum of item scores and represents difference between child's chronological age and age at which 90% of children in normative sample pass the items in that subscale.A higher derived score on a subscale indicates better performance on items in that subscale relative to other children of same age who have taken the test.Among subscales,Personal-Social subscale ranges from -16 months to 24 months;others range from - 12 months to 24 months.All subscales have a population mean of 0 and a standard deviation of 3.
Time Frame: Week 8 through Week 32
Population: ITT Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Ganaxolone
Number analyzed (Participants) | 34
Scores on a scale
  Week 8 - Personal Social | -0.72 (3.899)
  Week 8 - Fine Motor-Adaptive | -1.56 (3.131)
  Week 8 - Language | -1.45 (2.798)
  Week 8 - Gross Motor | -1.05 (2.285)
  Week 20- Personal Social | -2.82 (6.081)
  Week 20- Fine Motor-Adaptive | -3.73 (5.123)
  Week 20- Language | -2.39 (5.615)
  Week 20 - Gross Motor | -2.69 (3.584)
  Week 32-Personal Social: number analyzed (Participants) | 26
  Week 32-Personal Social | -4.86 (5.659)
  Week 32-Fine Motor-Adaptive: number analyzed (Participants) | 26
  Week 32-Fine Motor-Adaptive | -6.80 (4.952)
  Week 32-Language: number analyzed (Participants) | 26
  Week 32-Language | -6.58 (4.336)
  Week 32-Gross Motor: number analyzed (Participants) | 26
  Week 32-Gross Motor | -6.13 (4.509)

9. Secondary Outcome: Percentage of Total Spasm-free Days and Cumulative Spasm-free Days as Determined From the Seizure Diary.
Description: Percentage of total spasm-free days during a visit period is defined as total number of spasm free days as recorded in the Seizure Diary/ total number of days during that period, multiplied by 100.
  Percentage of cumulative total spasm-free days during a visit period is defined as sum of total number of spasm-free days during this period as recorded in the Seizure Diary/ total number of days in the treatment period, multiplied by 100.
Time Frame: Weeks 4 through Week 32
Population: ITT Population. Only those participants with data available at the indicated time point were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of Days
Arm/Group | Ganaxolone
Number analyzed (Participants) | 45
Percentage of Days
  Total Spasm-free days during Week 4 visit: number analyzed (Participants) | 43
  Total Spasm-free days during Week 4 visit | 11.10 (23.657)
  Total Spasm-free days during Week 8 visit: number analyzed (Participants) | 37
  Total Spasm-free days during Week 8 visit | 18.74 (32.654)
  Total Spasm-free days during Week 14 visit: number analyzed (Participants) | 36
  Total Spasm-free days during Week 14 visit | 20.74 (34.817)
  Total Spasm-free days during Week 20 visit: number analyzed (Participants) | 34
  Total Spasm-free days during Week 20 visit | 28.79 (40.163)
  Total Spasm-free days during Week 26 visit: number analyzed (Participants) | 30
  Total Spasm-free days during Week 26 visit | 28.73 (39.711)
  Total Spasm-free days during week 32 visit: number analyzed (Participants) | 26
  Total Spasm-free days during week 32 visit | 27.99 (39.259)
  Cumulative Spasm-free days during Week 4 visit | 10.86 (20.374)
  Cumulative Spasm-free days during Week 8 visit: number analyzed (Participants) | 40
  Cumulative Spasm-free days during Week 8 visit | 13.82 (23.433)
  Cumulative Spasm-free days during Week 14 visit: number analyzed (Participants) | 38
  Cumulative Spasm-free days during Week 14 visit | 15.70 (25.769)
  Cumulative Spasm-free days during Week 20 visit: number analyzed (Participants) | 36
  Cumulative Spasm-free days during Week 20 visit | 19.97 (28.501)
  Cumulative Spasm-free days during Week 26 visit: number analyzed (Participants) | 32
  Cumulative Spasm-free days during Week 26 visit | 22.07 (31.105)
  Cumulative Spasm-free days during Week 32 visit: number analyzed (Participants) | 27
  Cumulative Spasm-free days during Week 32 visit | 22.99 (30.140)

ADVERSE EVENTS:
Time Frame: Up to Week 32
Description: AEs and SAEs were collected in ITT Population. No separate analysis was performed to report results by doses.
Arm/Group | Ganaxolone
All-Cause Mortality (participants affected / at risk) | 2/54
Serious Adverse Events (participants affected / at risk) | 24/54
Other Adverse Events (participants affected / at risk) | 47/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ganaxolone (N=54)
Infantile spasms (Nervous system disorders) | 5
Convulsion (Nervous system disorders) | 4
Pyrexia (General disorders) | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3
Epilepsy (Nervous system disorders) | 2
Gastroenteritis (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Failure to thrive (Metabolism and nutrition disorders) | 2
Oral intake reduced (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ganaxolone (N=54)
Pyrexia (General disorders) | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 19
Upper respiratory tract infection (Infections and infestations) | 18
Vomiting (Gastrointestinal disorders) | 15
Nasopharyngitis (Infections and infestations) | 13
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11
Convulsion (Nervous system disorders) | 9
Urinary tract infection (Infections and infestations) | 8
Diarrhea (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 7
Teething (Gastrointestinal disorders) | 7
Somnolence (Nervous system disorders) | 7
Gastroesophageal reflux disease (Gastrointestinal disorders) | 6
Irritability (General disorders) | 6
Infantile spasms (Nervous system disorders) | 6
Ear infection (Infections and infestations) | 5
Influenza (Infections and infestations) | 5
Rhinitis (Infections and infestations) | 5
Dehydration (Metabolism and nutrition disorders) | 5
Tonic convulsion (Nervous system disorders) | 4
Oral intake reduced (Metabolism and nutrition disorders) | 4
Insomnia (Psychiatric disorders) | 4
Bronchitis (Infections and infestations) | 3
Gastroenteritis (Infections and infestations) | 3
Otitis media (Infections and infestations) | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3
Lethargy (Nervous system disorders) | 3
Metabolic acidosis (Metabolism and nutrition disorders) | 3
Hemoglobin decreased (Investigations) | 3
Anemia (Blood and lymphatic system disorders) | 3

LIMITATIONS AND CAVEATS:
Seizure-free information is not available

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No